CLINICAL TRIAL: NCT04251598
Title: Effect of the "I am Protecting my Child From the Sun" Program Based on Social Cognitive Theory, on Parent Behaviors
Brief Title: I am Protecting my Child From the Sun Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Adem SÜMEN, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TDK-2018-3501
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Skin Neoplasms; Parents; Behavior and Behavior Mechanisms; Child Behavior; Health Behavior
Keywords: Skin Cancer; Sun Protection; Parent Behavior; Social Cognitive Theory; Public Health Nursing
MeSH Terms: conditions — Skin Neoplasms; Behavior; Child Behavior; Health Behavior | interventions — Spermine Synthase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Education group (Experimental): Only "I am Protecting my Child From the Sun" program was given.
  Interventions: Behavioral: I Am Protecting My Child from the Sun
- Education + SMS group (Experimental): The "I am Protecting my Child From the Sun" program was given. After the program, an SMS message was sent on Wednesday and Saturday for 12 weeks. A total of 25 SMS messages were sent to remind the subject and applications.
  Interventions: Behavioral: I Am Protecting My Child from the Sun; Behavioral: SMS for sun protection
- Control group (No Intervention): No attempt was made by the researcher during the study. Only data collection was carried out. At the end of the research, the "I am Protecting my Child From the Sun" program was given..

INTERVENTIONS:
Behavioral: I Am Protecting My Child from the Sun — The parents in the intervention group were administered the "I Am Protecting My Child from the Sun" program for a period of six weeks.
  Intervention groups received Sun Protection Guide for Parents, Developmental, Characteristics of 3-6 Age Group Children Brochure, Melanoma Brochure, Video, Frame, Key chain, Magnet, Puzzle, Sunscreen product, T-shirt, hat and UV testing wristband.
  Arms: Education + SMS group; Education group
Behavioral: SMS for sun protection — While the education+SMS group, in addition to the program, also received a total of 25 short text messages twice a week.
  Arms: Education + SMS group

SUMMARY:
This study aimed to examine the effect of the "I Am Protecting My Child from the Sun" program, based on social cognitive theory, on parents' sun-protection product use and sun avoidance behaviors. The "I Am Protecting My Child from the Sun" program, based on Social Cognitive Theory, and the sending of short reminder messages had positive effects on the parents' behaviors related to protecting themselves and their children from the sun.

DETAILED DESCRIPTION:
This study aimed to examine the effect of the "I Am Protecting My Child from the Sun" program, based on social cognitive theory, on parents' sun-protection product use and sun avoidance behaviors. Organized as a randomized controlled experimental study conducted on three groups with a pre- and post-test follow-up design, the study was carried out in Manavgat between April 2018 and October 2018 and included the participation of 185 parents, of which 63 were in the education group, 62 were in the education+SMS group, and 60 were in the control group. The parents in the intervention group were administered the "I Am Protecting My Child from the Sun" program for a period of six weeks, while the education+SMS group, in addition to the program, also received a total of 25 short text messages twice a week. Data were collected using the Parent Information Form, Skin Cancer Risk Perception Form, Skin Cancer and Sun Knowledge Scale, Parental Self-Efficacy Scale, Parental Sun Protection Scales, and Parent Behaviors Regarding Protecting Themselves and Their Children from The Sun Question Form.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Being least literate
* No communication problems in terms of hearing, seeing and understanding
* Being a mobile phone user to receive text messages sent by the researcher
* Living in the same home with the child
* Joining both parents or one of the parents
* No possibility of leaving the region during the research

Exclusion Criteria:

* Skin cancer diagnosis / history
* Having a family history of skin cancer

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Parental Sun Protection Scales | 9 months
  The Self-Efficacy of the Use of Sunscreen Products consists of 5 items, Norms/Attitudes for the Use of Sunscreen Products consists of 6 items, Expectancies for the Use of Sunscreen Products consists of 6 items and Impediments to the Use of Sunscreen Products consists of 3 items in products; The Self - Efficacy of Sun Avoidance consists of 5 items, Norms/Attitudes for Sun Avoidance consists of 4 items, Tanning Expectancies consists of 4 items and Expectancies for Sun Avoidance consists of 5 items in Parental Sun Protection Scales. To calculate the scores of the scale, the items are numbered from 1 to 5. Each subscale will be evaluated within itself in the scales and it is expected that the scales of Impediments to the Use of Sunscreen Products and Tanning Expectancies scales have low scores and the other scales have high scores.
Sun Protection Applications of Parents for Themselves and Child's | 9 months
  The questionnaire is prepared according to the literature and consists of Sun Protection Applications of Parents for Themselves and Sun Protection Applications of Parents for Child's sections and five questions. It questions the sun protection practices for sunscreen, long-sleeved clothing, hat, sunglasses and shade. Answers to questions range from "never", " sometimes" and "always".

SECONDARY OUTCOMES:
Skin Cancer and Sun Knowledge Scale | 9 months
  The Skin Cancer and Sun Knowledge Scale consists of 25 items and evaluates information about five fields: the indications of sun protection, suntanning, skin cancer risk factors, prevention of skin cancer, and skin cancer. The items consist of 15 correct-incorrect and 10 multiple-choice questions. For each item, correct answers are symbolized by (1) and incorrect by (0). Total points are 0-25 on the scale. The higher the score obtained, the higher the knowledge level.
Skin Cancer Risk Perception | 9 months
  In the Skin Cancer Risk Perception questionnaire, there is a question that questions parents' risk of developing skin cancer, and two questions that question the possibility of developing skin cancer over the next 10 years and their lives. Parents' skin cancer risk perception was grouped between "very low" and "very high" and evaluated between 1 and 10 points, respectively. The increase in the score obtained is interpreted as high risk perception.
Parental Competence Scale | 9 months
  Parental Competence Scale consists of 11 items and one dimension to evaluate parents' parenting skills. The lowest 11 points and the highest 77 points can be obtained from the scale.
Skin Self-Examination | 9 months
  Skin self-examination practices were obtained by asking.

CONTACTS AND LOCATIONS:
Overall Officials: Selma Öncel, PhD, RN, Professor, Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Kumluca Faculty of Health Sciences, Antalya, Kumluca, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
I want to share "I am Protecting my Child From the Sun" program protocol with other researchers.
Supporting Information: Study Protocol, CSR
Time Frame: The study is completed
Access Criteria: After the study is published as an article

REFERENCES:
- [Derived] Sumen A, Oncel S. The effect of 'I am Protecting my Child from the Sun' programme on parental sun protection behaviours: Randomized controlled trial. J Adv Nurs. 2021 Jan;77(1):387-400. doi: 10.1111/jan.14614. Epub 2020 Oct 22. PMID 33089943